CLINICAL TRIAL: NCT03894137
Title: The Acute Effect of Grains of Paradise (Aframomum Melegueta) on Resting Energy Expenditure in Lean, Healthy, Adults
Brief Title: The Acute Effect of Grains of Paradise (Aframomum Melegueta) on REE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Plexus Worldwide (Industry)
Collaborators: George Mason University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 1355504-1
Record Dates: First submitted 2019-03-25; First posted 2019-03-28 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Obesity
Keywords: Grains of Paradise; energy metabolism; substrate oxidation
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Grains of Paradise (Experimental)
  Interventions: Dietary Supplement: Grains of Paradise (Aframomum Melegueta)
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Grains of Paradise (Aframomum Melegueta)

INTERVENTIONS:
Dietary Supplement: Grains of Paradise (Aframomum Melegueta) — This is a randomized, double blind, crossover design testing the effect of grains of paradise on resting energy metabolism

SUMMARY:
Grains of paradise (Aframomumu melegueta) (GP), also known as Guinea pepper or Alligator pepper, belongs to the Zingiberaceae family, which is native to West Africa. GP seeds are used as a spice and also have wide-ranging ethnobotanical uses. GP seeds are very rich in non-volatile pungent compounds such as 6-paradol, 6-gingerol, 6-shogaol and related compounds. This feature may equip them with the power to activate the Sympathetic Nervous System and thereby increase EE, which has been demonstrated in rodents. Research suggest that ingestion of GP extract can result in sustained elevation of EE and a consequent reduction in body fat. Thus, there is some evidence that GP may have a potential thermogenic effect that could be useful as part of a weight loss treatment. However, there is no information on whether GP has the potential of improving and prolonging the thermogenic effects of bioactives known to elevate fatty acid mobilization and subsequent fat oxidation. This proposal will fill a void in the literature by testing for the first time in healthy, normal weight, human volunteers whether the ingestion of GP in combination with a commercially available complex containing caffeine, green tea, and forskolin has an enhanced acute effect on REE, the largest and most stable component of EE, as well as the ratio of fat:carbohydrate oxidation. This project will provide pilot data to support larger studies such as prospective studies and studies to compare the thermogenic effect with currently available compounds.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-65 years
* Men and women
* Able to provide written consent in English
* A body mass index between 18.5 and 30 kg/m2

Exclusion Criteria:

* Current smoker
* Claustrophobia
* Use of any prescribed or over-the-counter medication affecting metabolism
* Suffering from cardiac, hepatic, renal, pulmonary, endocrine or hematological disease
* Currently pregnant or breastfeeding
* Consuming more than 300mg of caffeine per day
* Consuming more than 2 alcoholic beverages per day.
* Performing more than 3 hrs/week of strenuous exercise
* Weight loss of more than 5% of body weight over the past 6 months
* Not willing to abstain from alcohol, caffeine and exercise for 24hr before each test day.
* Suffering from heartburn or a sensitivity to pungent compounds in foods

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Resting metabolic Rate (Liters of oxygen consumed per minute) | 3 weeks
  Metabolic cart (metabolic gas exchange, indirect calorimitry)

SECONDARY OUTCOMES:
Resting substrate oxidation | 3 weeks
  Metabolic cart (respiratory exchange ratio)

OTHER OUTCOMES:
Heart Rate (beats per minute) | 3 weeks
  pulse frequency over time
Blood Pressure (mmHg) | 3 weeks
  automatic blood pressure cuff